CLINICAL TRIAL: NCT03873025
Title: Phase Ib/II Trial of Histone Deacetylase Inhibitor CXD101 in Combination With Programmed Cell Death Protein-1 Inhibitor Pembrolizumab for Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Study of CXD101 in Combination With Pembrolizumab for Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: PLACARD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: There are insufficent funds to open the trial and start recruiting patients due to the impact of the COVID-19 pandemic.
Sponsor: University College, London (Other)
Collaborators: Celleron Therapeutics Ltd. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/17/0920
Record Dates: First submitted 2019-03-05; First posted 2019-03-13 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and CXD101 (Experimental): Initial dose ('dose level 0'):-
  Single 200mg pembrolizumab IV infusion (day 1) in combination with oral CXD101 20mg twice daily PO (days 1 to 5) given in 21-day cycles for 2 years or until termination of treatment due to disease progression or unacceptable toxicity.
  Reduced dose level ('Dose level -1'; if >1 DLT observed at dose level 0):
  Single 200mg pembrolizumab IV infusion (day 1) in combination with oral CXD101 given twice daily, 20mg in the morning and 10mg in the evening (days 1 to 5) given in 21-day cycles for 2 years or until termination of treatment due to disease progression or unacceptable toxicity.
  Interventions: Combination Product: Pembrolizumab and CXD101

INTERVENTIONS:
Combination Product: Pembrolizumab and CXD101 — Pembrolizumab is a humanised monoclonal antibody which targets the programmed cell death 1 (PD-1) receptor. It blocks a protective mechanism on cancer cells, and allow the immune system to destroy these cancer cells. CXD101 is a histone deacetylase (HDAC) inhibitor which kills cancer cells by blocking the vital functions of HDAC enzymes.

SUMMARY:
Trial Subjects (patients), will receive single infusions of pembrolizumab in combination with CXD101 every 3 weeks for two years or until disease progression or unacceptable toxicity develops.

DETAILED DESCRIPTION:
Trial Subjects (patients) who are deemed eligible for the trial will initially be entered into the safety run-in stage of the trial. Up to 12 patients will be registered into the safety run-in stage, in cohorts of 3 patients at a time.

3 patients will be registered initially and will be administered a single infusion of pembrolizumab (200mg, day 1) in combination with CXD101 (20mg twice daily days 1 to 5). This is dose level 0.

If 0 to 1 dose limiting toxicity (DLT) is observed, 3 more patients will be entered into the trial and treated at dose level 0. If 0 to 1 DLT is observed across all 6 patients, the maximum tolerated dose (MTD) will be declared and the expansion stage of the trial will be opened.

If more than 1 DLT is observed at dose level 0, 3 patients will be recruited and treated at dose level -1. The CXD101 dose will be reduced by 25% (20mg in the morning and 10mg in the evening, days 1 to 5), while the pembrolizumab dose will remain the same (200mg, day 1).

If 0 or 1 DLT is observed, 3 more patients will be recruited and treated at dose level -1. If 0 or 1 DLT is observed across all 6 patients the maximum tolerated dose will be declared and the expansion stage of the trial will be opened.

If more than 1 DLT is observed at dose level -1 the combination will be deemed excessively toxic and no further patients enrolled.

Once the MTD is declared, the cohort will be expanded and a further 33 patients will be treated at this dose level.

Patients will continue to receive pembrolizumab and CXD101 at 3 weekly intervals for a maximum of 2 years or until disease progression or unacceptable toxicity develops. Patients on pembrolizumab will be seen every 3 weeks during trial treatment. Patients who progress will be seen annually for disease status. Patients completing treating or who stop treatment early for reasons other than disease progression will be followed every 3 months for up to one year after the end of treatment, and annually thereafter until end of trial is declared (when the last patient has completed 1 year follow up).

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed DLBCL, relapsed/ refractory after ≥2 lines of prior therapy and not fit for ASCT or relapsed post ASCT. Eligible histologies include (a) diffuse large B-cell lymphoma NOS, (b) transformed indolent non-Hodgkin lymphoma (including Richter's transformation), (c) EBV positive DLBCL NOS, (d) high grade B-cell lymphoma with MYC and BCL2 and/or BCL6 translocations, (e) high grade B-cell lymphoma NOS & (f) primary mediastinal B-cell lymphoma
2. Measurable disease (of >15mm in a node or >10mm in extranodal tissue)
3. Age 18 years or over
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Adequate organ and bone marrow function: Hb >80g/L, neutrophils >1.0x10^9/L and platelets >75x10^9/L (without platelet transfusion support)
6. International normalised ratio (INR) or prothrombin time (PT) or Activated partial thromboplastin time (aPTT): ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
7. Adequate renal function: estimated creatinine clearance >60ml/min as calculated using the Cockroft-Gault equation
8. Adequate liver function, including:

   1. Bilirubin ≤1.5 x upper limit of normal (ULN).
   2. Aspartate or alanine transferase (AST or ALT) ≤2.5 x ULN
9. Negative serum or urine pregnancy test for women of childbearing potential (WOCBP)
10. Willing to comply with the contraceptive requirements of the trial
11. Written informed consent

Exclusion Criteria:

1. Post-transplant lymphoproliferative disorder
2. Women who are pregnant or breast feeding, or males expecting to conceive or father children at any point from the start of study treatment until 4 months after the last administration of study treatment
3. Patients with corrected QTc (QTcF or QTcB) interval >450msec
4. Clinically significant cardiac or respiratory disease:

   1. Cardiac disease: Myocardial infarction, severe/unstable angina pectoris within 6 months prior to starting study treatment, NYHA class III-IV heart failure
   2. Pulmonary disease causing ≥ grade 2 dyspnoea or patient requiring oxygen
5. Known involvement of the central nervous system with lymphoma
6. Clinically significant active infection requiring antibiotic or antiretroviral therapy
7. Active autoimmune disease that has required systemic treatment in the past 2 years
8. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
9. History of immune hepatitis or myocarditis
10. Systemic anti-cancer therapy within 4 weeks prior to starting study treatment (12 weeks for CAR T-cells)
11. Prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids and not have had radiation pneumonitis.
12. Received a live vaccine within 30 days prior to starting study treatment
13. Have taken an IMP/investigational device within 4 weeks prior to starting study treatment
14. Major surgery within 4 weeks prior to starting study treatment
15. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX 40, CD137)
16. Prior allogeneic haematopoietic stem cell transplant, solid organ allogeneic transplant or allogeneic CAR T-cell therapy. Prior use of autologous CAR T-cell therapy is allowed but patient must be ≥ 12 weeks post infusion prior to starting study treatment
17. Diagnosis of prior immunodeficiency or organ-transplant requiring immunosuppressive therapy, or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
18. Positive serology for hepatitis B or C unless (as) hepatitis B positive due to vaccination (HBsAb positive, all other tests negative) or (b) past hepatitis B infection with low risk of reactivation (HBsAb positive & HBcAb positive, other tests (including hepatitis B DNA) negative - PI/co-investigator approval needed
19. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients and/or a history of allergies to the excipients for CXD101
20. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
22. Non-haematological malignancy within the past 3 years with the exception of (a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer (b) carcinoma in situ of the cervix or breast, (c) prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels; or (d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study such as localised transitional cell carcinoma of the bladder or benign tumours of the adrenal gland or pancreas
23. Current or prior use of immunosuppressive therapy within 7 days prior to start of treatment except the following: intranasal, inhaled, topical steroids or local steroid injections (eg. Intra-articular injection); systemic corticosteroids at physiologic doses (<10mg/day or less of prednisolone or equivalent)
24. Patient unable to swallow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Safety run in: Determine the maximum tolerated dose of CXD101 given in combination with pembrolizumab | During first cycle of CXD101 + pembrolizumab (each cycle lasts 21 days; assessment will take into account dose limiting toxicities reported at any time during the first 21 days of treatment)
  MTD to be defined as the highest dose level where 0 or 1 Dose limiting toxicity is observed in 6 patients
Best Objective Response Rate | From baseline to end of cycle 6 of treatment (approximately 18 weeks; each cycle lasts 21 days)
  Proportion of patients achieving CR or PR during the first 6 cycles of CXD101 in combination with pembrolizumab using the RECIL criteria

SECONDARY OUTCOMES:
Overall Response Rate at the end of 4 cycles | From baseline to end of cycle 4 of treatment (approximately 12 weeks; each cycle lasts 21 days)
  Overall Response of the combination of CXD101 and Pembrolizumab
Response Duration | From start of treatment to time of disease progression (any time during study participation, minimum 3 years)
  Time from date of first response confirmation to the first date of progressive disease confirmation
Best Overall Response at any time point | From baseline to end of treatment (up to 2 years)
  Best Overall Response of CXD101 in combination with Pembrolizumab
Best response at end of cycle 6 of treatment | From baseline to end of cycle 6 of treatment (approximately 18 weeks; each cycle lasts 21 days)
  CR, PR, MR, Stable Disease, Progressive Disease rates over 6 weeks of treatment
Progression Free Survival | 52 weeks after commencement of CXD101 and Pembrolizumab
  Progression Free Survival at 1 year
Overall Survival | 52 weeks after commencement of CXD101 and Pembrolizumab
  Overall survival at 1 year
Incidence of treatment-emergent adverse events (safety and tolerability) | From start of CXD101 and Pembrolizumab until 5 months post-treatment
  Adverse events to be reported during and after treatment, coded using CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Graham Collins, Principal Investigator — Oxford University Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No